CLINICAL TRIAL: NCT00757185
Title: Compromised Microcirculation in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0801003437; R21HL093450 (NIH)
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: skin blood flow; microcirculation
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — ganirelix; Methyltestosterone

ARMS (2):
- 1 (Experimental): GNRH antagonist alone
  Interventions: Drug: ganirelix acetate
- 2 (Experimental): GnRH with Testosterone
  Interventions: Drug: methyl testosterone

INTERVENTIONS:
Drug: ganirelix acetate — GnRH antagonist, subcutaneous injection, 0.25 mg/day for 21 days
  Other Names: Antagon
  Arms: 1
Drug: methyl testosterone — testosterone, oral administration, day 5 of GnRH administration, 2.5 mg/day
  Arms: 2

SUMMARY:
The scientific aims of the study are to determine how peripheral microcirculatory responsiveness is altered in obese women with Polycystic Ovary Syndrome (PCOS) during local heating and to determine the mechanism for testosterone effects on peripheral microcirculatory responsiveness in women with PCOS.

DETAILED DESCRIPTION:
In these studies, we propose to use the skin as a relatively non-invasive model to examine cardiovascular and endothelial function in obese women with and without PCOS. Data have indicated an important role for testosterone in influencing the peripheral microcirculation. While testosterone can lead to vasodilation in the peripheral microcirculation in both men and in women without PCOS, testosterone appears to induce vasoconstriction in women with PCOS. The differential response between women with and without PCOS, and between men and women may be the result of differential ET-1 actions in the vessel, and regulated by the receptor subtype is involved in these actions.

ELIGIBILITY:
Inclusion Criteria:

* Obese women (18-35) years with and without PCOS

Exclusion Criteria:

* Conditions that would preclude safe use of hormones

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-02; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Skin blood flow and cutaneous vascular conductance | 6 non consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Nina Stachenfeld, PhD, Principal Investigator — John B. Pierce Laboratory
Locations (1):
- John B. Pierce Laboratory, New Haven, Connecticut, United States